CLINICAL TRIAL: NCT06529341
Title: Efficacy of High-precision Transcranial Direct Current Stimulation on Anxiety Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chun Wang, professor, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 123201004258009355
Record Dates: First submitted 2024-07-06; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Anxiety Disorders; High-definition Transcranial Direct Current Stimulation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-definition transcranial direct current stimulation (Experimental): HD-tDCS stimulated AD left OFC (2 mA, 20 minutes, cathode electrode placed in the Fp 1 area, and the remaining four positive electrodes placed AF3, AF7, Afz, Fpz, forming a circular 41 focused electric field mode for stimulation, twice a day, 20 minutes interval for 5 days)
  Interventions: Other: High-definition transcranial direct current stimulation
- High-definition transcranial direct current stimulation pseudo-stimulation control group (Active Comparator): The treatment parameters of the electrode were the same as the test group, the stimulation current rose to the same 2 mA current in the test group within 30 seconds, and the pre-stimulation for 1 minute, then gradually to 0 mA.
  Interventions: Other: High-definition transcranial direct current stimulation pseudo-stimulation control group

INTERVENTIONS:
Other: High-definition transcranial direct current stimulation — HD-tDCS stimulated AD left OFC (2 mA, 20 minutes, cathode electrode placed in the Fp 1 area, and the remaining four positive electrodes placed AF3, AF7, Afz, Fpz, forming a circular 41 focused electric field mode for stimulation, twice a day, 20 minutes interval for 5 days)
  Arms: High-definition transcranial direct current stimulation
Other: High-definition transcranial direct current stimulation pseudo-stimulation control group — The treatment parameters of the electrode were the same as the test group, the stimulation current rose to the same 2 mA current in the test group within 30 seconds, and the pre-stimulation for 1 minute, then gradually to 0 mA.
  Arms: High-definition transcranial direct current stimulation pseudo-stimulation control group

SUMMARY:
1. Current research has found that tDCS has a positive effect on improving the negative attention bias of AD patients, and this study uses HD-tDCS intervention to improve the cognitive function and neural mechanisms of AD patients in the OFC to provide a theoretical basis for AD neural mechanism research. Verify Hypothesis 1: HD-tDCS cathodal stimulation of the left OFC reduces the excitability of this region, modulates its connectivity with the attentional function network, and thus changes the emotional experience of social threat.
2. Currently, there is no consensus on the stimulation parameters for tDCS in the treatment of AD, and more evidence is needed to prove and explore. It is hoped that the HD-tDCS intervention protocol will become an effective treatment method for improving cognitive function and clinical symptoms in AD patients. Hypothesis 2: The HD-tDCS with intensified stimulation parameters (2mA, twice a day, with a 20-minute interval, for 5 consecutive days) has an impact on the main and secondary clinical variables of AD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the DSM-5 AD diagnostic criteria;
2. The Chinese version of the Brief International Neuropsychiatric Interview (MINI) screening meets the diagnosis;
3. Age: 18-55 years old;
4. The patient participated voluntarily, obtained the consent of the family members, and signed the informed consent form;
5. Scale score criteria: 14 points on the Hamilton Anxiety Scale (HAMA) and 17 points on the Hamilton Depression Scale (HAMD).

Exclusion Criteria:

1. Neurological diseases or other psychiatric disorders;
2. severe somatic diseases;
3. received medical treatment including medication, psychotherapy, electroconvulsive therapy, and physical therapy within the first half months of enrollment;
4. tDCS examination contraindications, such as intracranial metal or electronic implants, skull plate, or other skull implants.
5. Pregnancy and lactation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Scale | 1 week
  HAMA was assessed at baseline and late 5 days after treatment by a professionally trained physician (non-trial intervention) to understand the effectiveness of treatment. Clinical efficacy evaluation criteria: 75% was recovered, 50% was significant, 25% was effective, and <25% was invalid.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No